CLINICAL TRIAL: NCT00965731
Title: Phase 1/2, Open Label, Randomized Study Of The Safety, Efficacy, And Pharmacokinetics Of Erlotinib With Or Without Pf 02341066 In Patients With Advanced Non Small Cell Adenocarcinoma Of The Lung.
Brief Title: Erlotinib Is Being Studied With Or Without An Investigational Drug, PF-02341066, In Patients With Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A8081002; 2009-012377-35 (EudraCT Number)
Record Dates: First submitted 2009-08-24; First posted 2009-08-26 (Estimated); Results first posted 2013-01-14 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Lung Neoplasms; Crizotinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Erlotinib Hydrochloride; Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Erlotinib (Active Comparator)
  Interventions: Drug: Erlotinib
- Erlotinib + PF-02341066 (Experimental)
  Interventions: Drug: Erlotinib; Drug: PF-02341066

INTERVENTIONS:
Drug: Erlotinib — Erlotinib, 150 mg, QD will be administered orally on a continuous schedule (Phase 2 only)
  Arms: Erlotinib
Drug: Erlotinib — For Phase 1 - escalating doses of erlotinib will be administered orally on a continuous schedule. The planned doses to be evaluated are 100 and 150 mg QD. The dose determined in Phase 1 will be used in Phase 2
  Arms: Erlotinib + PF-02341066
Drug: PF-02341066 — For Phase 1 - escalating doses of PF-02341066 will be administered orally on a continuous schedule. The planned doses to be evaluated are 200 and 250 mg BID. The dose determined in Phase 1 will be used in Phase 2
  Arms: Erlotinib + PF-02341066

SUMMARY:
This is a Phase 1/2 study comparing the safety and anti-tumor activity of erlotinib alone versus erlotinib in combination with PF-02341066 in patients with advanced non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven diagnosis of Non-Small Cell Lung Cancer (NSCLC) that is locally advanced or metastatic and of the adenocarcinoma subtype (including mixed adenosquamous histology)
* evident disease progression by Response Evaluation Criterion in Solid Tumors (RECIST) after at least one but no more than 2 chemotherapy regimens for advanced disease
* tumors must have measurable disease as per RECIST

Exclusion Criteria:

* known interstitial lung disease
* prior treatment with an agent that is known or proposed to be active by action on EGFR tyrosine kinase or c-Met/HGF (Phase 2 Portion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (15):
- United States (15):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, Irvine Medical Center Pharmacy, Orange, California
  - University of California, Irving - Medical Center, Orange, California
  - University of California Irvin, Orange, California
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Siteman Cancer Center, City of Saint Peters, Missouri
  - Siteman Cancer Center -West County, Creve Coeur, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University, School of Medicine, St Louis, Missouri
  - OSU East, Columbus, Ohio
  - The Ohio State University James Cancer Hospital, Columbus, Ohio
  - James Care in Kenny, Columbus, Ohio
  - Cancer Therapy & Research Center @ UTHSCSA, San Antonio, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8081002&StudyName=Erlotinib%20Is%20Being%20Studied%20With%20Or%20Without%20An%20Investigational%20Drug%2C%20PF-02341066%2C%20In%20Patients%20With%20Lung%20Cancer

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was planned to include 2 phases; phase 1 was a dose escalation safety and pharmacokinetic (PK) study followed by a randomized phase 2 efficacy and safety study. The study was discontinued and phase 2 not started; no participants were enrolled in that phase of the study.
Groups:
- PF-02341066 (200 mg) and Erlotinib (100 mg): PF-02341066 200 milligrams (mg) administered orally twice daily (BID) in combination with erlotinib 100 mg administered orally once daily (QD) in a continuous schedule for 28 days (Cycle 1) and then in continuous 21-day cycles. Prior to combination treatment, participants completed a 7 to 14 day lead-in period where they received erlotinib 100 mg administered orally QD.
- PF-02341066 (150 mg) and Erlotinib (100 mg): PF-02341066 150 mg administered orally BID in combination with erlotinib 100 mg administered orally QD in a continuous schedule for 28 days (Cycle 1) and then in continuous 21-day cycles. Prior to combination treatment, participants completed a 7 to 14 day lead-in period where they received erlotinib 100 mg administered orally QD.
Period: Overall Study
Arm/Group | PF-02341066 (200 mg) and Erlotinib (100 mg) | PF-02341066 (150 mg) and Erlotinib (100 mg)
Started | 7 | 20 (Dose level given only after lower dose was successfully administered)
Completed | 0 | 0
Not Completed | 7 | 20
Not completed — Death | 0 | 4
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Other | 7 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-02341066 (200 mg) and Erlotinib (100 mg) | PF-02341066 (150 mg) and Erlotinib (100 mg) | Total
Number analyzed (Participants) | 7 | 20 | 27
Age, Customized [Number; unit: participants]
  18 to 44 years | 1 | 0 | 1
  45 to 64 years | 5 | 11 | 16
  greater than or equal to (≥) 65 | 1 | 9 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 13 | 19
  Male | 1 | 7 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLT) (Phase 1)
Description: Phase 1, first cycle DLT includes Grade (Gr) ≥4 hematologic possible drug-related toxicities and Gr ≥3 possible drug-related febrile neutropenia. Gr ≥3 non-hematological possible drug-related toxicities (except asymptomatic lab value elevation). Gr 3/4 nausea, vomiting or diarrhea. Gr 3 hypertension considered DLT if event unmanageable by approved pharmacologic agents or symptomatic sequelae despite medical intervention. Diagnosis of interstitial lung disease. Inability to deliver at least 80 percent (%) of planned dose during cycle 1 due to possible drug-related adverse events (AEs).
Time Frame: Baseline up to Day 28
Population: DLT evaluable population: all participants in dose escalation phase receiving at least 1 dose of study medication who did not have a major treatment deviation during the first cycle (for example, less than 80% of planned dose of PF-02341066 or erlotinib in cycle 1 for reasons other than treatment-related toxicities)
Measure: Number; unit: participants
Groups:
- PF-02341066 (200 mg) and Erlotinib (100 mg): PF-02341066 200 milligrams (mg) administered orally twice daily (BID) and erlotinib 100 mg administered orally once daily (QD) in a continuous schedule for 28 days (Cycle 1) and then in continuous 21-day cycles. Prior to combination treatment, participants completed a 7 to 14 day lead-in period where they received erlotinib 100 mg administered orally QD.
- PF-02341066 (150 mg) and Erlotinib (100 mg): PF-02341066 150 mg administered orally BID and erlotinib 100 mg administered orally QD in a continuous schedule for 28 days (Cycle 1) and then in continuous 21-day cycles. Prior to combination treatment, participants completed a 7 to 14 day lead-in period where they received erlotinib 100 mg administered orally QD.
Arm/Group | PF-02341066 (200 mg) and Erlotinib (100 mg) | PF-02341066 (150 mg) and Erlotinib (100 mg)
Number analyzed (Participants) | 6 | 16
participants | 2 | 3

2. Primary Outcome: Progression-Free Survival (Phase 2)
Description: Time in weeks from phase 2 study randomization to first documentation of objective disease progression or death due to any cause. Progression-Free Survival was calculated as (first event date minus randomization date plus 1) divided by 7.02. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD]), or from AE data (where the outcome was "Death"; date of death reported in notice of death was used).
Time Frame: Baseline, every 42 days up to 20 months, disease progression, or unacceptable toxicity
Population: Not analyzed due to phase 2 study termination
Groups:
- PF-02341066 and Erlotinib: PF-02341066 (BID) and erlotinib (QD) administered at the recommended Phase 2 dose (RP2D) in continuous 21-day cycles.
- Erlotinib: Erlotinib 150 mg was to be administered orally QD in continuous 21-day cycles
Arm/Group | PF-02341066 and Erlotinib | Erlotinib
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: PF-02341066 (Crizotinib) Area Under the Concentration-Time Curve During Dosing Interval (AUCtau) (Phase 1)
Description: AUCtau is a measure of the plasma exposure to PF-02341066. In this study, it is used to characterize PF-02341066 exposure after a single dose (Cycle 1 Day 1) and multiple doses (Cycle1 Day 15) of PF-02341066 were administered in combination of Erlotinib.
Time Frame: Cycle 1 (C1) Day 1 (D1) i.e., 1 day of giving crizotinib and erlotinib; and C1D15, i.e., 15 days of giving crizotinib and erlotinib
Population: Pharmacokinetic (PK) parameter analysis population included all participants in safety analysis set 1 who had at least 1 of the PK parameters of interest. Number of participants analyzed section in below table includes number of participants in PK analysis population. N=number of participants in treatment group contributing to summary statistics.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-02341066 (200 mg) and Erlotinib (100 mg) | PF-02341066 (150 mg) and Erlotinib (100 mg)
Number analyzed (Participants) | 7 | 19
ng*hr/mL
  C1D1 Crizotinib (N=7, 19) | 581.9 (49) | 400.3 (40)
  C1D15 Crizotinib (N=5, 14) | 2274 (43) | 1720 (40)

4. Secondary Outcome: PF-02341066 (Crizotinib) Maximum Observed Plasma Concentration (Cmax) (Phase 1)
Description: Cmax is a measure of the plasma exposure to PF-02341066. In this study, it is used to characterize PF-02341066 exposure after a single dose (Cycle 1 Day 1) and multiple doses (Cycle 1 Day 15) of PF-02341066 were administered in combination of Erlotinib
Time Frame: C1D1 i.e., 1 day of giving crizotinib and erlotinib; and C1D15, i.e., 15 days of giving crizotinib and erlotinib
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-02341066 (200 mg) and Erlotinib (100 mg) | PF-02341066 (150 mg) and Erlotinib (100 mg)
Number analyzed (Participants) | 7 | 19
ng/mL
  C1D1 Crizotinib (N=7, 19) | 86.75 (37) | 65.31 (50)
  C1D15 Crizotinib (N=5, 14) | 251.0 (46) | 185.9 (40)

5. Secondary Outcome: PF-02341066 (Crizotinib) Apparent Oral Clearance (CL/F) (Phase 1)
Description: Apparent oral Clearance is a measure of combination of the rate at which a drug is removed from the blood (CL) and the bioavailability (F) after oral dose. In this study, It is used to characterize PF-02341066 CL/F after multiple doses (Cycle 1 Day 15) of PF-02341066 were administered in combination of Erlotinib.
Time Frame: C1D15 i.e., 15 days of giving crizotinib and erlotinib
Population: The pharmacokinetic (PK) parameter analysis population was defined as all participants in the safety analysis set 1 who had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | PF-02341066 (200 mg) and Erlotinib (100 mg) | PF-02341066 (150 mg) and Erlotinib (100 mg)
Number analyzed (Participants) | 5 | 14
L/hr | 88.02 (43) | 87.20 (40)

6. Secondary Outcome: PF-06260182 Area Under the Concentration-Time Curve During Dosing Interval (AUCtau) (Phase 1)
Description: AUCtau is a measure of the plasma exposure to PF-06260182, a PF-02341066 metabolite. In this study, it is used to characterize the metabolite exposure after a single dose (Cycle 1 Day 1) and multiple doses (Cycle 1 Day 15) of PF-02341066 were administered in combination of Erlotinib.
Time Frame: C1D1 i.e., 1 day of giving crizotinib and erlotinib; and C1D15, i.e., 15 days of giving crizotinib and erlotinib
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-02341066 (200 mg) and Erlotinib (100 mg) | PF-02341066 (150 mg) and Erlotinib (100 mg)
Number analyzed (Participants) | 7 | 19
ng*hr/mL
  C1D1 PF-06260182 (N=7, 19) | 16.48 (58) | 14.03 (72)
  C1D15 PF-06260182 (N=5, 14) | 60.36 (63) | 57.77 (66)

7. Secondary Outcome: PF-06260182 Maximum Observed Plasma Concentration (Cmax) (Phase 1)
Description: Cmax is a measure of the plasma exposure to PF-06260182, a PF-02341066 metabolite. In this study, it is used to characterize the metabolite exposure after a single dose (Cycle 1 Day 1) and multiple doses (Cycle 1 Day 15) of PF-02341066 were administered in combination of Erlotinib.
Time Frame: C1D1 i.e., 1 day of giving crizotinib and erlotinib; and C1D15, i.e., 15 days of giving crizotinib and erlotinib
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-02341066 (200 mg) and Erlotinib (100 mg) | PF-02341066 (150 mg) and Erlotinib (100 mg)
Number analyzed (Participants) | 7 | 19
ng/mL
  C1D1 PF-06260182 (N=7, 19) | 2.625 (49) | 2.087 (63)
  C1D15 PF-06260182 (N=5, 14) | 7.093 (54) | 6.508 (63)

8. Secondary Outcome: Molecular Weight Adjusted PF-06260182-to-PF-02341006 Ratio of AUCtau (Phase 1)
Description: Molecular weight adjusted PF-06260182-to-PF-02341006 ratio of AUCtau is a measure of how much PF-02341066 (parent drug) was converted to the metabolite PF-06260182 after PF-02341066 dosing. In this study, it is used to characterize the metabolite-to-parent ratio exposure after a single dose (Cycle 1 Day 1) and multiple doses (Cycle 1 Day 15) of PF-02341066 were administered in combination of Erlotinib.
Time Frame: C1D1 i.e., 1 day of giving crizotinib and erlotinib; and C1D15, i.e., 15 days of giving crizotinib and erlotinib
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | PF-02341066 (200 mg) and Erlotinib (100 mg) | PF-02341066 (150 mg) and Erlotinib (100 mg)
Number analyzed (Participants) | 7 | 19
Ratio
  C1D1 (N=7, 19) | 0.02748 (23) | 0.03395 (45)
  C1D15 (N=5, 14) | 0.02574 (27) | 0.03258 (31)

9. Secondary Outcome: Erlotinib Area Under the Concentration-Time Curve During Dosing Interval (AUCtau) (Phase 1)
Description: AUCtau is a measure of the plasma exposure to erlotinib. In this study, it is used to characterize erlotinib exposure after multiple doses of erlotinib were administered alone (Day -1) and in combination of PF-02341066 (Cycle 1 Day 1 and Day 15).
Time Frame: C1D-1 i.e., 1 day prior to initiation of continuous dosing of crizotinib; C1D1 i.e., 1 day of giving crizotinib and erlotinib; and C1D15, i.e., 15 days of giving crizotinib and erlotinib
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-02341066 (200 mg) and Erlotinib (100 mg) | PF-02341066 (150 mg) and Erlotinib (100 mg)
Number analyzed (Participants) | 7 | 19
ng*hr/mL
  C1D-1 Erlotinib Alone (N=7,19) | 23490 (31) | 26880 (39)
  C1D1 Erlotinib+Crizotinib Single Dose (N=7,19) | 26520 (25) | 30040 (39)
  C1D15 Erlotinib+Crizotinib Multiple Doses (N=5,14) | 41770 (27) | 38910 (49)

10. Secondary Outcome: Erlotinib Maximum Observed Plasma Concentration (Cmax) (Phase 1)
Description: Cmax is a measure of the plasma exposure to erlotinib. In this study, it is used to characterize erlotinib exposure after multiple doses of erlotinib were administered alone (Day -1) and in combination of PF-02341066 (Cycle 1 Day 1 and Day 15).
Time Frame: as for outcome 9
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-02341066 (200 mg) and Erlotinib (100 mg) | PF-02341066 (150 mg) and Erlotinib (100 mg)
Number analyzed (Participants) | 7 | 19
ng/mL
  C1D-1 Erlotinib Alone (N=7,19) | 1593 (26) | 1797 (36)
  C1D1 Erlotinib+Crizotinib Single Dose (N=7,19) | 1452 (21) | 1723 (38)
  C1D15 Erlotinib+Crizotinib Multiple Doses (N=5,14) | 2546 (24) | 2346 (43)

11. Secondary Outcome: Erlotinib Apparent Oral Clearance (CL/F) (Phase 1)
Description: Apparent oral Clearance is a measure of combination of the rate at which a drug is removed from the blood (CL) and the bioavailability (F) after oral dose. In this study, it is used to characterize erlotinib CL/F after multiple doses in combination with PF-02341066 (Cycle 1 Day 15).
Time Frame: C1D15 i.e., 15 days of giving crizotinib and erlotinib
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | PF-02341066 (200 mg) and Erlotinib (100 mg) | PF-02341066 (150 mg) and Erlotinib (100 mg)
Number analyzed (Participants) | 5 | 14
L/hr | 2.395 (27) | 2.572 (49)

12. Secondary Outcome: Ratio of Adjusted Means of Erlotinib AUCtau (Crizotinib + Erlotinib / Erlotinib Alone) (Phase 1)
Description: Ratio of adjusted means of Erlotinib AUCtau (Crizotinib + Erlotinib / Erlotinib Alone) is a measure of the plasma exposure to erlotinib after erlotinib dosing with crizotinib compared with that after erlotinib dosing alone. In this study, it is used to characterize the effect magnitude of crizotinib on the erlotinib exposure after combinational use of crizotinib and erlotinib.
Time Frame: C1D-1 (i.e., 1 day prior to initiation of continuous dosing of crizotinib) to C1D15 (i.e., 15 days of giving crizotinib and erlotinib)
Population: The PK parameter analysis population was defined as all participants in the safety analysis set 1 who had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio in percentage
Arm/Group | PF-02341066 (200 mg) and Erlotinib (100 mg) | PF-02341066 (150 mg) and Erlotinib (100 mg)
Number analyzed (Participants) | 7 | 19
Ratio in percentage | 184.80 (40) [149.67 to 228.18] | 149.41 (43) [125.87 to 177.36]

13. Secondary Outcome: Ratio of Adjusted Means of Erlotinib Cmax (Crizotinib + Erlotinib / Erlotinib Alone) (Phase 1)
Description: Ratio of adjusted means of Erlotinib Cmax (Crizotinib + Erlotinib / Erlotinib Alone) is a measure of the plasma exposure to erlotinib after erlotinib dosing with crizotinib compared with that after erlotinib dosing alone. In this study, it is used to characterize the effect magnitude of crizotinib on the erlotinib exposure after combinational use of crizotinib and erlotinib.
Time Frame: as for outcome 12
Population: as for outcome 5
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio in percentage
Arm/Group | PF-02341066 (200 mg) and Erlotinib (100 mg) | PF-02341066 (150 mg) and Erlotinib (100 mg)
Number analyzed (Participants) | 7 | 19
Ratio in percentage | 160.15 (49) [121.06 to 211.86] | 134.60 (27) [115.23 to 157.22]

14. Secondary Outcome: Progression-Free Survival (Phase 1)
Description: Time in weeks from phase 1 randomization to first documentation of objective disease progression or death due to any cause. Progression-Free Survival was calculated as (first event date minus randomization date plus 1) divided by 7.02. Tumor progression was determined from oncologic assessment data (where data meet the criteria for PD), or from AE data (where the outcome was "Death"; date of death reported in notice of death was used).
Time Frame: Baseline, every 42 days until disease progression or unacceptable toxicity
Population: not analyzed due to small number of study participants
Arm/Group | PF-02341066 (200 mg) and Erlotinib (100 mg) | PF-02341066 (150 mg) and Erlotinib (100 mg)
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Duration of Response (Phase 1)
Description: Median duration (50 percent [%]) of tumor response. Duration of response (DR) defined as time from start of first documented objective tumor response [Complete Response (CR) or Partial Response (PR)] to first documented objective tumor progression or death due to any cause, whichever occurs first. DR calculated as (Weeks) = (the end date for DR minus first subsequent confirmed CR or PR plus 1) divided by 7.02. CR: disappearance of a target lesions. PR: at least 30% decrease in the sum of diameters of target lesions.
Time Frame: Baseline, every 42 days until disease progression or unacceptable toxicity
Population: not analyzed due to small number of responses
Arm/Group | PF-02341066 (200 mg) and Erlotinib (100 mg) | PF-02341066 (150 mg) and Erlotinib (100 mg)
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Percentage of Participants With Objective Response (Phase 1)
Description: Percentage of participants during phase 1 with objective response based assessment of confirmed CR or confirmed PR according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1). Confirmed responses: persist on repeat imaging study at least 4 weeks after initial documentation of response. CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). No new lesions and disappearance of all non-target lesions. PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of nontarget disease. No new lesions.
Time Frame: Baseline, every 42 days until disease progression or unacceptable toxicity
Population: Response Evaluable Population: all participants enrolled into the Phase 1 portion of the study who receive at least one dose of study medication (either PF-02341066 or erlotinib) and have an adequate baseline tumor assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-02341066 (200 mg) and Erlotinib (100 mg) | PF-02341066 (150 mg) and Erlotinib (100 mg)
Number analyzed (Participants) | 7 | 18
percentage of participants | 14.3 [0.4 to 57.9] | 5.6 [0.1 to 27.3]

17. Secondary Outcome: Plasma Level of Soluble Marker: c-Met Ectodomain (Phase 1)
Description: Levels of soluble protein biomarker c-MET was analyzed at Baseline and at Day 50.
Time Frame: Baseline and Day 50 (Cycle 3, Day 1)
Population: The soluble biomarker evaluable population was defined as participants from the safety analysis set of phase 1 who had a soluble protein blood sample taken prior to dosing on Cycle 3 Day 1 and 1 soluble biomarker evaluation after dosing on Cycle 3 Day 1.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-02341066 (200 mg) and Erlotinib (100 mg) | PF-02341066 (150 mg) and Erlotinib (100 mg)
Number analyzed (Participants) | 1 | 7
nanogram per milliliter (ng/mL)
  Baseline | 1560.0 (NA) — Not available as there is only one participant. | 1454.6 (303.93)
  C3D1 0 Hour | 1870.0 (NA) — Not available as there is only one participant. | 1525.9 (442.01)
  C3D1 6 Hour | 1660.0 (NA) — Not available as there is only one participant. | 1600.0 (369.05)

18. Secondary Outcome: Plasma Level of Soluble Marker: Hepatocyte Growth Factor (HGF) Scatter Factor (Phase 1)
Time Frame: Baseline and Day 50 (Cycle 3, Day 1)
Population: Plasma level of soluble marker HGF scatter factor not analyzed due to prior experience with high levels of intra participant variability
Arm/Group | PF-02341066 (200 mg) and Erlotinib (100 mg) | PF-02341066 (150 mg) and Erlotinib (100 mg)
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Plasma Level of Soluble Marker: c-Met Ectodomain (Phase 2)
Time Frame: Baseline and Day 50 (Cycle 3, Day 1)
Population: Not analyzed due to phase 2 study termination
Arm/Group | PF-02341066 and Erlotinib | Erlotinib
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Plasma Level of Soluble Marker: HGF Scatter Factor (Phase 2)
Time Frame: Baseline and Day 50 (Cycle 3, Day 1)
Population: Not analyzed due to phase 2 study termination
Arm/Group | PF-02341066 and Erlotinib | Erlotinib
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Duration of Response (Phase 2)
Description: Median duration (50%) of tumor response. DR defined as time from start of first documented objective tumor response (CR or PR) to first documented objective tumor progression or death due to any cause, whichever occurs first. DR calculated as (Weeks) = (the end date for DR minus first subsequent confirmed CR or PR plus 1) divided by 7.02. CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). No new lesions and disappearance of all non-target lesions. PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of nontarget disease. No new lesions.
Time Frame: Baseline, every 42 days up to 20 months, disease progression, or unacceptable toxicity
Population: Not analyzed due to phase 2 study termination
Arm/Group | PF-02341066 and Erlotinib | Erlotinib
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Percentage of Participants With Confirmed CR, PR or Stable Disease (SD) at Phase 2
Description: Percentage of participants during phase 2 with confirmed CR, confirmed PR or SD according to RECIST 1.1. Also known as Disease Control Rate (DCR). CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). No new lesions and disappearance of all non-target lesions. PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of nontarget disease. No new lesions. SD: neither sufficient shrinkage or increase to qualify for PR or PD.
Time Frame: Week 6 and Week 12
Population: Not analyzed due to phase 2 study termination
Arm/Group | PF-02341066 and Erlotinib | Erlotinib
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Percentage of Participants With Objective Response (Phase 2)
Description: Percentage of participants during phase 2 with objective response based assessment of confirmed CR or confirmed PR according to RECIST (1.1). Confirmed responses: persist on repeat imaging study at least 4 weeks after initial documentation of response. CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). No new lesions and disappearance of all non-target lesions. PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of nontarget disease. No new lesions.
Time Frame: Baseline, every 42 days up to 20 months, disease progression, or unacceptable toxicity
Population: Not analyzed due to phase 2 study termination
Arm/Group | PF-02341066 and Erlotinib | Erlotinib
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Overall Survival (OS) at Phase 2
Description: Time in months from randomization to date of death due to any cause. OS was calculated as (the death date minus the date of randomization plus 1) divided by 30.4.
Time Frame: Baseline until death, up to 20 months
Population: Not analyzed due to phase 2 study termination
Arm/Group | PF-02341066 and Erlotinib | Erlotinib
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: European Organization for Research and Treatment of Cancer (EORTC), Quality of Life Questionnaire (QLQ-C30) Score at Phase 2
Description: Phase 2 EORTC QLQ-C30: included functional scales (physical, role, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting) and single items (dyspnoea, appetite loss, insomnia, constipation/diarrhea and financial difficulties). Most questions used 4 point scale (1 'Not at all' to 4 'Very much'; 2 questions used 7-point scale (1 'very poor' to 7 'Excellent'). Scores averaged, transformed to 0-100 scale; higher score=better level of functioning or greater degree of symptoms.
Time Frame: Baseline and every 21 days, up to 20 months
Population: Not analyzed due to phase 2 study termination
Arm/Group | PF-02341066 and Erlotinib | Erlotinib
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: EORTC Quality of Life Questionnaire -Lung Cancer 13 (QLQ-LC13) Score at Phase 2
Description: QLQ-LC13 consisted of 13 questions relating to disease symptoms specific to lung cancer and treatment side effects typical of treatment with chemotherapy and radiotherapy. The 13 questions comprised 1 multi-item scale for dyspnea and 10 single-item symptoms and side effects (coughing, hemoptysis, sore mouth, dysphagia, neuropathy, alopecia, and medicine for pain). Recall period: past week; response range: not at all to very much. Scale score range: 0 to 100. Higher symptom score = greater degree of symptoms.
Time Frame: Baseline and every 21 days, up to 20 months
Population: Not analyzed due to phase 2 study termination
Arm/Group | PF-02341066 and Erlotinib | Erlotinib
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Plasma Concentration of PF-02341066 and Erlotinib (Phase 2)
Description: Plasma concentration of PF-02341066 and erlotinib when administered in combination during phase 2
Time Frame: Day 1 of cycles 1, 3, and 5 (i.e., up to 15 weeks) at 0 (pre-dose) and 2 to 6 hours post dose
Population: Not analyzed due to phase 2 study termination
Arm/Group | PF-02341066 and Erlotinib | Erlotinib
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Plasma Concentration of Erlotinib (Phase 2)
Description: Plasma concentration of erlotinib when administered as a single agent during phase 2
Time Frame: Day 1 of cycles 1, 3, and 5 (i.e., up to 15 weeks) at 0 hours (pre-dose)
Population: Not analyzed due to phase 2 study termination
Arm/Group | PF-02341066 and Erlotinib | Erlotinib
Number analyzed (Participants) | 0 | 0

29. Secondary Outcome: Percentage of Participants With Mutations in Tumor Tissue (Phase 2)
Description: Tumor tissue samples collected for molecular profiling were to be analyzed to assess Kirsten rat sarcoma (KRAS) mutations, mutations, amplification and expression of Epidermal Growth Factor Receptor (EGFR) and c-Met, and echinoderm microtubule-associated protein-like 4-anaplastic large cell receptor kinase (EML4-ALK) fusion in tumors.
Time Frame: Screening
Population: Not analyzed due to phase 2 study termination
Groups:
- PF-02341066 and Erlotinib: PF-02341033 (BID) and erlotinib (QD) administered at the recommended Phase 2 dose (RP2D) in continuous 21-day cycles
Arm/Group | PF-02341066 and Erlotinib | Erlotinib
Number analyzed (Participants) | 0 | 0

30. Other Pre Specified Outcome: Maximum Tolerated Dose (MTD) of PF-02341066 When Administered in Combination With Erlotinib (Phase 1)
Description: MTD: the combination dose level of PF-02341066 and erlotinib in which 0/6 or 1/6 participants experienced DLT after 28 days of treatment (Cycle 1) with the next higher dose level having at least 2/3 or 2/6 participants with DLT during Cycle 1 of treatment.
Time Frame: Baseline up to 28 days (Cycle 1)
Population: DLT evaluable population
Measure: Number; unit: mg
Groups:
- All Treated Participants (Phase 1): All participants who received PF-02341066 (200 mg or 150 mg) administered orally BID and erlotinib 100 mg administered orally QD in a continuous schedule for 28 days (Cycle 1) and then in continuous 21-day cycles. Prior to combination treatment, participants completed a 7 to 14 day lead-in period where they received erlotinib 100 mg administered orally QD.
Arm/Group | All Treated Participants (Phase 1)
Number analyzed (Participants) | 22
mg
  PF-02341066 (BID) | 150
  Erlotinib (QD) | 100

31. Other Pre Specified Outcome: Recommended Phase 2 Dose (RP2D) of PF-02341066 When Administered in Combination With Erlotinib (Phase 1)
Description: If no more than 1/6 participants presented with a DLT during Cycle 1 at the MTD, then this dose level was considered the RP2D. If >1/6 participants experienced a DLT, then the previous lower level was considered the MTD and RP2D.
Time Frame: Baseline up to 28 days (Cycle 1)
Population: DLT evaluable population
Measure: Number; unit: mg
Arm/Group | All Treated Participants (Phase 1)
Number analyzed (Participants) | 22
mg
  PF-02341066 (BID) | 150
  Erlotinib (QD) | 100

ADVERSE EVENTS:
Time Frame: Up to 28 days after the last dose of study treatment (up to approximately 20 months)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-02341066 (200 mg) and Erlotinib (100 mg) | PF-02341066 (150 mg) and Erlotinib (100 mg)
Serious Adverse Events (participants affected / at risk) | 2/7 | 8/20
Other Adverse Events (participants affected / at risk) | 7/7 | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-02341066 (200 mg) and Erlotinib (100 mg) (N=7) | PF-02341066 (150 mg) and Erlotinib (100 mg) (N=20)
Disease progression (General disorders) | 0 | 4
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2
Viral infection (Infections and infestations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-02341066 (200 mg) and Erlotinib (100 mg) (N=7) | PF-02341066 (150 mg) and Erlotinib (100 mg) (N=20)
Anaemia (Blood and lymphatic system disorders) | 1 | 3
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Adrenal disorder (Endocrine disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 1
Dry eye (Eye disorders) | 1 | 0
Eye pruritus (Eye disorders) | 1 | 1
Eyelid pain (Eye disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 1 | 0
Photopsia (Eye disorders) | 0 | 1
Scotoma (Eye disorders) | 1 | 1
Trichiasis (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 3
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3
Constipation (Gastrointestinal disorders) | 0 | 5
Diarrhoea (Gastrointestinal disorders) | 6 | 16
Dyspepsia (Gastrointestinal disorders) | 1 | 3
Dysphagia (Gastrointestinal disorders) | 1 | 2
Flatulence (Gastrointestinal disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 11
Oesophageal pain (Gastrointestinal disorders) | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 2
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 8
Asthenia (General disorders) | 0 | 2
Catheter site swelling (General disorders) | 0 | 1
Chest discomfort (General disorders) | 0 | 1
Chills (General disorders) | 0 | 2
Fatigue (General disorders) | 3 | 14
Malaise (General disorders) | 1 | 1
Mucosal inflammation (General disorders) | 0 | 3
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 1
Pain (General disorders) | 2 | 0
Pyrexia (General disorders) | 1 | 3
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0
Abscess (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Rash pustular (Infections and infestations) | 2 | 0
Rhinitis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 2
Blood alkaline phosphatase decreased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 2
Blood creatinine increased (Investigations) | 1 | 0
Breath sounds abnormal (Investigations) | 1 | 2
Breath sounds absent (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 3
White blood cell count decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 12
Dehydration (Metabolism and nutrition disorders) | 1 | 4
Fluid retention (Metabolism and nutrition disorders) | 0 | 1
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Ataxia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2
Dysgeusia (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 1
Hyperaesthesia (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Vocal cord paralysis (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 4
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 13
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 2
Phlebitis superficial (Vascular disorders) | 1 | 0
Nail bed infection (Infections and infestations) | 1 | 0
Local swelling (General disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The sponsor terminated phase 2 of this study; no data was collected during phase 2, leading to phase 2 outcomes not analyzed. The decision was based on strategic considerations regarding the clinical program only; there were no safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.